CLINICAL TRIAL: NCT02475330
Title: Phase II Trial of Flaxseed to Prevent Pneumonopathy After Chemoradiation for Lung Cancer
Brief Title: Dietary Flaxseed in NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patient compliance
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Supportive Care
Other Study IDs: UPCC 28514
Record Dates: First submitted 2015-06-16; First posted 2015-06-18 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dietary Supplement: Flaxseed (Experimental)
  Interventions: Dietary Supplement: Flaxseed

INTERVENTIONS:
Dietary Supplement: Flaxseed — Whole grain flaxseed diet consisting of 40g flaxseed ingested per day

SUMMARY:
This single arm Phase II trial will investigate the feasibility of dietary flaxseed (FS) supplementation in subjects receiving definitive chemoradiotherapy for non-small cell lung cancer (NSCLC). Subjects will ingest FS for a period of approximately 8 to 9 weeks during the course of radiation treatment. Study participation and surveillance will last approximately 6 months. Subject specimen collection will include: blood, urine, and buccal swabs at 5 time points.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 18 and older
* Current diagnosis of non-small cell lung cancer (NSCLC) including patients who have metastatic disease requiring definitive thoracic and mediastinal radiotherapy with concurrent chemotherapy.
* Able to provide written informed consent and comply with all study procedures
* Total planned radiation dose to gross disease 60-70 Gy.

Exclusion Criteria:

* Current diagnosis of disease of the gastrointestinal system, liver, or kidneys which could result in altered metabolism or excretion of the study medication (history of major gastrointestinal tract surgery, gastrectomy, gastrostomy, bowel resection, etc.) or history of chronic gastrointestinal disorders (ulcerative colitis, regional enteritis, or gastrointestinal bleeding)
* Known hypersensitivity to flaxseed or any of its metabolites, or wheat products
* Taking or has taken an investigational drug within 14 days.
* Taking or has taken Amifostine or Mucomyst (N-acetylcysteine) within 14 days
* Current or prior use of flaxseed, flax-containing products, soybeans, or soy-containing products
* Current or prior use (limited to prior 14 days) of dietary supplements such as herbals or botanicals
* Prior thoracic and/or mediastinal radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Rate of Radiation-Induced Lung Injury | 6 months
  Rate of RILI after flaxseed administration in a population of patients receiving definitive chemoradiotherapy for lung cancer.
Rates of Grade >3 Radiation Pneumonitis | 6 months
  Toxicity and tolerability data of dietary FS administration during chemoradiotherapy

SECONDARY OUTCOMES:
Concentration of G-CSF | 6 months
Concentration of GM-CSF | 6 months
Concentration of IFN-α | 6 months
Concentration of IFN-γ | 6 months
Concentration of IL-1β | 6 months
Concentration of IL-1RA | 6 months
Concentration of IL-2 | 6 months
Concentration of IL-2R | 6 months
Concentration of IL-4 | 6 months
Concentration of IL-5 | 6 months
Concentration of IL-6 | 6 months
Concentration of IL-7 | 6 months
Concentration of IL-8 | 6 months
Concentration of IL-10 | 6 months
Concentration of IL-12 | 6 months
Concentration of IL-13 | 6 months
Concentration of IL-15 | 6 months
Concentration of IL-17 | 6 months
Concentration of TNF-α | 6 months
Concentration of Eotaxin | 6 months
Concentration of IP-10 | 6 months
Concentration of MCP-1 | 6 months
Concentration of MIG | 6 months
Concentration of MIP-1α | 6 months
Concentration of MIP-1ß | 6 months
Concentration of RANTES | 6 months
Concentration of EGF | 6 months
Concentration of FGF-Basic | 6 months
Concentration of HGF | 6 months
Concentration of VEGF | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Berman, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Lim TL, Pietrofesa RA, Arguiri E, Koumenis C, Feigenberg S, Simone CB 2nd, Rengan R, Cengel K, Levin WP, Christofidou-Solomidou M, Berman AT. Phase II Trial of Flaxseed to Prevent Acute Complications After Chemoradiation for Lung Cancer. J Altern Complement Med. 2021 Oct;27(10):824-831. doi: 10.1089/acm.2020.0542. Epub 2021 Jun 23. PMID 34161146

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT02475330/Prot_SAP_000.pdf